CLINICAL TRIAL: NCT04424927
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of PRV-015 in Adult Patients With Non-Responsive Celiac Disease as an Adjunct to a Gluten-free Diet
Brief Title: PRV-015 in Gluten-free Diet Non-responsive Celiac Disease
Acronym: PROACTIVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Provention Bio, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRV-015-002b; DRI18114 (Other: Sanofi Identifier); 2020-000649-16 (EudraCT Number)
Record Dates: First submitted 2020-05-28; First posted 2020-06-11 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PRV-015 Low Dose (Experimental): PRV-015 Low Dose, sterile solution for subcutaneous administration
  Interventions: Biological: PRV-015
- PRV-015 Medium Dose (Experimental): PRV-015 Medium Dose, sterile solution for subcutaneous administration
  Interventions: Biological: PRV-015
- PRV-015 High Dose (Experimental): PRV-015 High Dose, sterile solution for subcutaneous administration
  Interventions: Biological: PRV-015
- Placebo (Placebo Comparator): Placebo, sterile solution for subcutaneous administration
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: PRV-015 — Fully human monoclonal antibody against interleukin 15 (IL-15)
  Arms: PRV-015 High Dose; PRV-015 Low Dose; PRV-015 Medium Dose
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of PRV-015 in adult patients with non-responsive celiac disease (NRCD) who are on a gluten-free diet (GFD).

DETAILED DESCRIPTION:
PRV-015-002b is a Phase 2b, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy and safety of 3 dose regimens of PRV-015 in adult patients with NRCD who are on a GFD.

Eligible subjects include male or female adults, 18 to 70 years of age, with a diagnosis of celiac disease and have followed a GFD for at least 12 consecutive months, yet continue to experience symptoms.

Study drug (1 of the 3 doses of PRV-015 or placebo) will be administered in a double-blind fashion, followed by a safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of celiac disease by intestinal biopsy
* Following a GFD for at least 12 consecutive months
* Must have detectable (above the lower limit of detection) serum celiac-related antibodies
* Must have human leukocyte antigen DQ (HLA-DQ) typing consistent with celiac disease (DQ2 and/or DQ8)
* Subjects must have had at least one of the following symptoms at least once per week during the month before screening: diarrhea, loose stools, abdominal pain, abdominal cramping, bloating, or gas.
* Body weight between 35 and 120 kg

Exclusion Criteria:

* Current diagnosis of any severe complication of celiac disease, such as refractory celiac disease type 1 (RCD-I) or RCD-II, enteropathy-associated T-cell lymphoma (EATL), ulcerative jejunitis, or gastrointestinal (GI) perforation
* Diagnosis of any chronic, active GI disease other than celiac disease
* Presence of any active infection
* Selective immunoglobulin A (IgA) deficiency, defined as having undetectable levels of IgA
* Known or suspected exposure to coronavirus disease 2019 (COVID-19) infection in the 4 weeks before screening
* Administration of a live vaccine within 14 days prior to randomization and the first administration of study drug
* History or presence of any clinically significant disease that, in the opinion of the Investigator, may confound the subject's participation and follow-up in the clinical trial or put the subject at unnecessary risk
* Females who are pregnant or planning to become pregnant during the study period, or who are currently breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (36):
- United States (28):
  - Clinical Site, Los Angeles, California
  - Clinical Site, Ventura, California
  - Clinical Site, Denver, Colorado
  - Clinical Site, Leesburg, Florida
  - Clinical Site, Tampa, Florida
  - Clinical Site, Winter Park, Florida
  - Clinical Site, Chicago, Illinois
  - Clinical Trial Site, Northbrook, Illinois
  - Clinical Trial Site, Chevy Chase, Maryland
  - Clinical Site, Boston, Massachusetts
  - Clinical Site, Chesterfield, Michigan
  - Clinical Site, Rochester, Minnesota
  - Clinical Site, Morristown, New Jersey
  - Clinical Trial Site, Brooklyn, New York
  - Clinical Site, New Windsor, New York
  - Clinical Trial Site, New York, New York
  - Clinical Site, Raleigh, North Carolina
  - Clinical Trial Site, Dublin, Ohio
  - Clinical Site, Philadelphia, Pennsylvania
  - Clinical Site, Uniontown, Pennsylvania
  - Clinical Site, Warwick, Rhode Island
  - Clinical Trial Site, North Charleston, South Carolina
  - Clinical Site, Nashville, Tennessee
  - Clinical Trial Site, Cedar Park, Texas
  - Clinical Site, Garland, Texas
  - Clinical Site, West Jordan, Utah
  - Clinical Site, Bellevue, Washington
  - Clinical Site, Tacoma, Washington
- Clinical Site, Hamilton, Ontario, Canada
- Clinical Site, Amsterdam, Netherlands
- Spain (6):
  - Clinical Site, Seville, Andalusia
  - Clinical Site, León, Castille and León
  - Clinical Trial Site, Terrassa, Catalonia
  - Clinical Trial Site, Girona
  - Clinical Trial Site, Lleida
  - Clinical Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 39 centers in 4 countries. A total of 648 participants were screened between 24 August 2020 and 16 January 2024, of which 255 participants were screen failures and 5 participants discontinued before run-in period. Screen failures were mainly due to not meeting eligibility criteria.
Pre-assignment Details: A total of 388 participants entered the single-blind placebo run-in period and among them, 1 participant never received treatment and was not started after signing the ICF, 9 participants discontinued during run-in or were not dosed, and 27 participants were considered run-in failures. Another 126 participants were considered randomization failures. A total of 226 participants were enrolled and randomized in the study.
Groups:
- Single-blind: Placebo: Participants received placebo subcutaneous (SC) injection every 2 weeks (q2w) in single-blind placebo run-in period for 4 weeks.
- Double-blind: Placebo: Participants received placebo matching with PRV-015 SC injection q2w in double-blind treatment period for 24 weeks.
- Double-blind: PRV-015 100 mg: Participants received PRV-015 100 milligram (mg) SC injection q2w in double-blind treatment period for 24 weeks.
- Double-blind: PRV-015 300 mg: Participants received PRV-015 300 mg SC injection q2w in double-blind treatment period for 24 weeks.
- Double-blind: PRV-015 600 mg: Participants received PRV-015 600 mg SC injection q2w in double-blind treatment period for 24 weeks.
Period: Single-blind Period (4 Weeks)
Arm/Group | Single-blind: Placebo | Double-blind: Placebo | Double-blind: PRV-015 100 mg | Double-blind: PRV-015 300 mg | Double-blind: PRV-015 600 mg
Started | 388 | 0 | 0 | 0 | 0
Received Treatment | 387 | 0 | 0 | 0 | 0
Completed | 352 | 0 | 0 | 0 | 0
Not Completed | 36 | 0 | 0 | 0 | 0
Not completed — Not treated | 1 | 0 | 0 | 0 | 0
Not completed — Run-in failure | 27 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 0 | 0 | 0 | 0
Not completed — Investigator or sponsor judgement | 1 | 0 | 0 | 0 | 0
Period: Double-blind Period (24 Weeks)
Arm/Group | Single-blind: Placebo | Double-blind: Placebo | Double-blind: PRV-015 100 mg | Double-blind: PRV-015 300 mg | Double-blind: PRV-015 600 mg
Started | 0 (Only participants started in double-blind treatment period are reported.) | 57 (Only participants started in double-blind treatment period are reported.) | 56 (Only participants started in double-blind treatment period are reported.) | 57 (Only participants started in double-blind treatment period are reported.) | 56 (Only participants started in double-blind treatment period are reported.)
Received Treatment | 0 | 57 | 56 | 57 | 54
Completed | 0 | 51 | 47 | 51 | 49
Not Completed | 0 | 6 | 9 | 6 | 7
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 5 | 5 | 6
Not completed — Investigator or Sponsor judgement | 0 | 1 | 0 | 0 | 1
Not completed — Other | 0 | 1 | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Single-blind period: Participants treated with single-blind placebo in run-in period are included.
  Double-blind period: The intent-to-treat analysis set included all randomized participants.
Groups:
- Single-blind: Placebo: Participants received placebo SC injection q2w in single-blind placebo run-in period for 4 weeks.
- Double-blind: PRV-015 100 mg: Participants received PRV-015 100 mg SC injection q2w in double-blind treatment period for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Single-blind: Placebo | Double-blind: Placebo | Double-blind: PRV-015 100 mg | Double-blind: PRV-015 300 mg | Double-blind: PRV-015 600 mg | Total
Number analyzed (Participants) | 387 | 57 | 56 | 57 | 56 | 613
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Baseline measure data reported for each study period separately.
  years
    Single-blind period: number analyzed (Participants) | 387 | 0 | 0 | 0 | 0 | 387
    Single-blind period | 41.2 (13.8) |  |  |  |  | 41.2 (13.8)
    Double-blind period: number analyzed (Participants) | 0 | 57 | 56 | 57 | 56 | 226
    Double-blind period |  | 41.0 (14.53) | 41.9 (14.82) | 39.0 (12.25) | 37.9 (12.58) | 39.9 (13.59)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline measure data reported for each study period separately.
  Participants
    Single-blind period: number analyzed (Participants) | 387 | 0 | 0 | 0 | 0 | 387
    Single-blind period: Female | 313 | 0 | 0 | 0 | 0 | 313
    Single-blind period: Male | 74 | 0 | 0 | 0 | 0 | 74
    Double-blind period: number analyzed (Participants) | 0 | 57 | 56 | 57 | 56 | 226
    Double-blind period: Female | 0 | 53 | 38 | 50 | 45 | 186
    Double-blind period: Male | 0 | 4 | 18 | 7 | 11 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Baseline measure data reported for each study period separately.
  Participants
    Single-blind period: number analyzed (Participants) | 387 | 0 | 0 | 0 | 0 | 387
    Single-blind period: Black or African American | 4 |  |  |  |  | 4
    Single-blind period: White | 375 |  |  |  |  | 375
    Single-blind period: Asian | 1 |  |  |  |  | 1
    Single-blind period: American Indian or Alaska Native | 2 |  |  |  |  | 2
    Single-blind period: Not Reported | 3 |  |  |  |  | 3
    Single-blind period: Unknown | 1 |  |  |  |  | 1
    Single-blind period: Multiple | 1 |  |  |  |  | 1
    Double-blind period: number analyzed (Participants) | 0 | 57 | 56 | 57 | 56 | 226
    Double-blind period: Black or African American |  | 0 | 1 | 0 | 0 | 1
    Double-blind period: White |  | 57 | 55 | 56 | 53 | 221
    Double-blind period: Asian |  | 0 | 0 | 0 | 0 | 0
    Double-blind period: American Indian or Alaska Native |  | 0 | 0 | 0 | 0 | 0
    Double-blind period: Not Reported |  | 0 | 0 | 0 | 2 | 2
    Double-blind period: Unknown |  | 0 | 0 | 0 | 1 | 1
    Double-blind period: Multiple |  | 0 | 0 | 1 | 0 | 1
Celiac Disease Patient Reported Outcome (CeD PRO) Abdominal Symptoms Domain Score [Count of Participants; unit: Participants] — The CeD PRO questionnaire was captured daily in the electronic (e)Diary. The questionnaire included 9 items: abdominal cramping, abdominal pain, bloating, gas, diarrhea, loose stool, nausea, headache and tiredness. Participants were asked to rate their symptom severity on an 11-point scale and scores range from 0 (not experiencing the symptom) to 10 (the worst possible symptom experience). Abdominal Symptoms domain included abdominal cramping, abdominal pain, bloating and gas. Total score for abdominal symptoms domain range from 0 to 40. Higher scores indicated worse outcome. Population: Baseline measure data reported for each study period separately. Analysis was not performed during the single-blind placebo period for this measurement as it is specific to the double-blind periods and IMP per the protocol, and the single-blind number analyzed is 0.
  Participants
    Single-blind period: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
    Single-blind period: Score: <3 |  |  |  |  |  | 0
    Single-blind period: Score: >=3 |  |  |  |  |  | 0
    Double-blind period: number analyzed (Participants) | 0 | 57 | 56 | 57 | 56 | 226
    Double-blind period: Score: <3 |  | 13 | 13 | 13 | 13 | 52
    Double-blind period: Score: >=3 |  | 44 | 43 | 44 | 43 | 174
Number of Participants for Stratification Factor Villous Height-to-Crypt Depth Ratio (VH:CD) [Count of Participants; unit: Participants] — Esophagogastroduodenoscopy and biopsy were performed to determine villus height and crypt depth and their ratio. Population: Baseline measure data reported for each study period separately. Analysis was not performed during the single-blind placebo period for this measurement as it is specific to the double-blind periods and IMP per the protocol, and the single-blind number analyzed is 0.
  Participants
    Single-blind period: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
    Single-blind period: Ratio: <2 |  |  |  |  |  | 0
    Single-blind period: Ratio: >=2 |  |  |  |  |  | 0
    Double-blind period: number analyzed (Participants) | 0 | 57 | 56 | 57 | 56 | 226
    Double-blind period: Ratio: <2 |  | 37 | 37 | 37 | 36 | 147
    Double-blind period: Ratio: >=2 |  | 20 | 19 | 20 | 20 | 79

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Celiac Disease Patient-Reported Outcome Abdominal Symptoms Domain Score Through Week 24
Description: The CeD PRO questionnaire was captured daily in the eDiary. The questionnaire included 9 items: abdominal cramping, abdominal pain, bloating, gas, diarrhea, loose stool, nausea, headache and tiredness. Participants were asked to rate their symptom severity on an 11-point scale and scores range from 0 (not experiencing the symptom) to 10 (the worst possible symptom experience). Abdominal Symptoms domain included abdominal cramping, abdominal pain, bloating and gas. Total score for abdominal symptoms domain range from 0 to 40. Higher scores indicated worse outcome. Baseline abdominal symptoms domain score was defined as the average of the daily scores for the last week of the placebo run-in period.
Time Frame: Baseline (average of Day -7 to Day -1) up to Week 24
Population: The modified intent-to-treat (mITT) analysis set included all randomized participants who received at least 1 dose of double-blind treatment. Only participants with data collected at baseline and up to Week 24 are reported.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Placebo: Participants received placebo matching with PRV-015 SC injection q2w in double-blind treatment period for 24 weeks.
- PRV-015 100 mg: Participants received PRV-015 100 mg SC injection q2w in double-blind treatment period for 24 weeks.
- PRV-015 300 mg: Participants received PRV-015 300 mg SC injection q2w in double-blind treatment period for 24 weeks.
- PRV-015 600 mg: Participants received PRV-015 600 mg SC injection q2w in double-blind treatment period for 24 weeks.
Arm/Group | Placebo | PRV-015 100 mg | PRV-015 300 mg | PRV-015 600 mg
Number analyzed (Participants) | 56 | 55 | 56 | 52
score on a scale | -1.32 [-1.66 to -0.98] | -1.28 [-1.62 to -0.94] | -1.21 [-1.55 to -0.88] | -1.28 [-1.63 to -0.93]
Statistical Analysis 1: Comparison: Placebo vs PRV-015 100 mg; Estimates/p-value are from a mixed model for repeated measures (MMRM) with treatment, week, and treatment by week as fixed effects; continuous baseline CeD PRO Abdominal Symptoms domain score and baseline VH:CD ratio as covariates, and participant as a random effect; Test type: Other; p = 0.8543, MMRM; Least square (LS) mean difference = 0.04, 95% CI 2-sided [-0.43 to 0.52]
Statistical Analysis 2: Comparison: Placebo vs PRV-015 300 mg; Estimates/p-value are from a MMRM with treatment, week, and treatment by week as fixed effects; continuous baseline CeD PRO Abdominal Symptoms domain score and baseline VH:CD ratio as covariates, and participant as a random effect; Test type: Other; p = 0.6552, MMRM; LS mean difference = 0.11, 95% CI 2-sided [-0.37 to 0.59]
Statistical Analysis 3: Comparison: Placebo vs PRV-015 600 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.8705, MMRM; LS mean difference = 0.04, 95% CI 2-sided [-0.45 to 0.53]

2. Secondary Outcome: Absolute Change From Baseline in Celiac Disease Patient-Reported Outcome Diarrhea and Loose Stool Domain Score Through Week 24
Description: The CeD PRO questionnaire was captured daily in the eDiary. The questionnaire included 9 items: abdominal cramping, abdominal pain, bloating, gas, diarrhea, loose stool, nausea, headache and tiredness. Participants were asked to rate their symptom severity on an 11-point scale and scores range from 0 (not experiencing the symptom) to 10 (the worst possible symptom experience). Diarrhea and loose stool domain included diarrhea and loose stool. Total score for diarrhea and loose stool domain range from 0 to 20. Higher scores indicated worse outcome. Baseline diarrhea and loose stool domain score was defined as the average of the daily scores for the last week of the placebo run-in period.
Time Frame: Baseline (average of Day -7 to Day -1) up to Week 24
Population: The mITT analysis set included all randomized participants who received at least 1 dose of double-blind treatment. Only participants with data collected at baseline and up to Week 24 are reported.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | PRV-015 100 mg | PRV-015 300 mg | PRV-015 600 mg
Number analyzed (Participants) | 56 | 55 | 56 | 52
score on a scale | -0.77 [-1.15 to -0.40] | -0.66 [-1.04 to -0.28] | -1.02 [-1.39 to -0.64] | -1.07 [-1.46 to -0.68]
Statistical Analysis 1: Comparison: Placebo vs PRV-015 100 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.6757, MMRM; LS mean difference = 0.11, 95% CI 2-sided [-0.42 to 0.65]
Statistical Analysis 2: Comparison: Placebo vs PRV-015 300 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.3645, MMRM; LS mean difference = -0.25, 95% CI 2-sided [-0.78 to 0.29]
Statistical Analysis 3: Comparison: Placebo vs PRV-015 600 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.2791, MMRM; LS mean difference = -0.30, 95% CI 2-sided [-0.84 to 0.24]

3. Secondary Outcome: Absolute Change From Baseline in Celiac Disease Patient-Reported Outcome Total Gastrointestinal (GI) Score Through Week 24
Description: The CeD PRO questionnaire was captured daily in the eDiary. The questionnaire included 9 items: abdominal cramping, abdominal pain, bloating, gas, diarrhea, loose stool, nausea, headache and tiredness. Participants were asked to rate their symptom severity on an 11-point scale and scores range from 0 (not experiencing the symptom) to 10 (the worst possible symptom experience). Total GI domain included abdominal symptoms domain, diarrhea, loose stool and nausea. Total GI score range from 0 to 70. Higher scores indicated worse outcome. Baseline GI score was defined as the average of the daily scores for the last week of the placebo run-in period.
Time Frame: Baseline (average of Day -7 to Day -1) up to Week 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | PRV-015 100 mg | PRV-015 300 mg | PRV-015 600 mg
Number analyzed (Participants) | 56 | 55 | 56 | 52
score on a scale | -0.89 [-1.15 to -0.63] | -0.84 [-1.10 to -0.57] | -0.88 [-1.14 to -0.62] | -1.05 [-1.32 to -0.78]
Statistical Analysis 1: Comparison: Placebo vs PRV-015 100 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.7829, MMRM; LS mean difference = 0.05, 95% CI 2-sided [-0.32 to 0.42]
Statistical Analysis 2: Comparison: Placebo vs PRV-015 300 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.9503, MMRM; LS mean difference = 0.01, 95% CI 2-sided [-0.36 to 0.38]
Statistical Analysis 3: Comparison: Placebo vs PRV-015 600 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.4107, MMRM; LS mean difference = -0.16, 95% CI 2-sided [-0.54 to 0.22]

4. Secondary Outcome: Absolute Change From Baseline in Intraepithelial Lymphocyte (IEL) Density at Week 24
Description: The small intestinal mucosal inflammation was measured by IEL density using immunohistochemistry. Baseline was defined as IEL density from the esophagogastroduodenoscopy biopsy conducted during the run-in period.
Time Frame: Baseline to Week 24
Population: The mITT analysis set included all randomized participants who received at least 1 dose of double-blind treatment. Only participants with data collected at baseline and Week 24 are reported.
Measure: Least Squares Mean (95% Confidence Interval); unit: cells/100 epithelial cells
Arm/Group | Placebo | PRV-015 100 mg | PRV-015 300 mg | PRV-015 600 mg
Number analyzed (Participants) | 51 | 49 | 51 | 48
cells/100 epithelial cells | -0.39 [-3.82 to 3.03] | 1.54 [-1.99 to 5.07] | -4.11 [-7.56 to -0.66] | -4.53 [-8.13 to -0.93]
Statistical Analysis 1: Comparison: Placebo vs PRV-015 100 mg; Estimates/p-value are from an analysis of covariance (ANCOVA) model with treatment as a fixed effect. Continuous baseline CeD PRO Abdominal Symptoms domain score and baseline VH:CD ratio are included as covariates; Test type: Other; p = 0.4397, ANCOVA; LS mean difference = 1.94, 95% CI 2-sided [-3.00 to 6.87]
Statistical Analysis 2: Comparison: Placebo vs PRV-015 300 mg; Estimates/p-value are from an ANCOVA model with treatment as a fixed effect. Continuous baseline CeD PRO Abdominal Symptoms domain score and baseline VH:CD ratio are included as covariates; Test type: Other; p = 0.1337, ANCOVA; LS mean difference = -3.72, 95% CI 2-sided [-8.58 to 1.15]
Statistical Analysis 3: Comparison: Placebo vs PRV-015 600 mg; [analysis description as in outcome 4, analysis 2]; Test type: Other; p = 0.1021, ANCOVA; LS mean difference = -4.14, 95% CI 2-sided [-9.11 to 0.83]

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (SAEs) and Treatment-Emergent Adverse Events of Special Interest (AESIs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug. An SAE was defined as any AE that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. AESIs included severe opportunistic infections and hypersensitivity reactions of at least moderate severity. A TEAE was defined as an AE that occurred from the first dose of post-randomization study drug administration through the end of the study.
Time Frame: From first dose of study drug administration (Day 1) up to 28 days after the last dose administration, 197 days
Population: The Safety analysis set included all participants who received at least 1 dose of the study drug post-randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PRV-015 100 mg | PRV-015 300 mg | PRV-015 600 mg
Number analyzed (Participants) | 57 | 56 | 57 | 54
Participants
  Any TEAE | 34 | 34 | 36 | 29
  TEAE leading to study treatment discontinuation | 1 | 1 | 2 | 0
  Treatment-emergent SAE | 1 | 0 | 0 | 1
  Treatment-emergent AESI | 2 | 1 | 1 | 1

6. Secondary Outcome: Number of Participants With Potentially Clinically Important Changes in Hematology
Description: Blood samples were collected to determine the hematology laboratory important changes. CHG= Change from baseline hemoglobin.
Time Frame: From first dose of study drug administration (Day 1) up to 28 days after the last dose administration, 197 days
Population: The Safety analysis set included all participants who received at least 1 dose of the study drug post-randomization. Only participants with data collected are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PRV-015 100 mg | PRV-015 300 mg | PRV-015 600 mg
Number analyzed (Participants) | 57 | 56 | 57 | 53
Participants
  Hemoglobin: CHG <=-20 g/L | 0 | 0 | 1 | 2
  Neutrophils: <1 10^9/L | 2 | 1 | 4 | 2

7. Secondary Outcome: Number of Participants With Potentially Clinically Important Changes in Clinical Chemistry
Description: Blood samples were collected to determine the clinical chemistry laboratory important changes. ULN= Upper limit of normal, mmol/L= millimoles per liter and mcmol/L= micromoles per liter.
Time Frame: From first dose of study drug administration (Day 1) up to 28 days after the last dose administration, 197 days
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PRV-015 100 mg | PRV-015 300 mg | PRV-015 600 mg
Number analyzed (Participants) | 57 | 56 | 57 | 53
Participants
  Alanine Aminotransferase: >=3x ULN | 1 | 4 | 1 | 2
  Aspartate Aminotransferase: >=3x ULN | 1 | 2 | 0 | 0
  Chloride: >125 mmol/L | 1 | 0 | 1 | 0
  Creatinine: >=132 mcmol/L | 1 | 1 | 0 | 0
  Potassium: >6 mmol/L | 0 | 0 | 2 | 1
  Sodium: <125 mmol/L | 0 | 0 | 1 | 0

8. Secondary Outcome: Number of Participants With Potentially Clinically Important Changes in Urinalysis
Description: Urine samples were collected to determine the important changes in urine. TNTC= Too numerous to count, LPF= Low power field and HPF= High power field.
Time Frame: From first dose of study drug administration (Day 1) up to 28 days after the last dose administration, 197 days
Population: The Safety analysis set included all participants who received at least 1 dose of the study drug post-randomization. Only participants with data collected for each specific parameter are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PRV-015 100 mg | PRV-015 300 mg | PRV-015 600 mg
Number analyzed (Participants) | 57 | 56 | 57 | 53
Participants
  Bacteria: Present: number analyzed (Participants) | 54 | 51 | 55 | 47
  Bacteria: Present | 54 | 51 | 55 | 47
  Crystals: Present: number analyzed (Participants) | 3 | 4 | 2 | 5
  Crystals: Present | 3 | 4 | 2 | 5
  Erythrocytes (/HPF): Many/TNTC: number analyzed (Participants) | 55 | 56 | 56 | 53
  Erythrocytes (/HPF): Many/TNTC | 1 | 0 | 4 | 3
  Glucose: 3+/4+ | 1 | 2 | 1 | 0
  Hyaline Casts (/HPF): Few/Moderate/Many: number analyzed (Participants) | 8 | 7 | 9 | 7
  Hyaline Casts (/HPF): Few/Moderate/Many | 3 | 2 | 3 | 0
  Hyaline Casts (/LPF): Few/Moderate/Many: number analyzed (Participants) | 0 | 2 | 1 | 0
  Hyaline Casts (/LPF): Few/Moderate/Many |  | 1 | 1 |
  Ketones: 3+ | 1 | 2 | 3 | 1
  Leukocyte Esterase: 3+/4+ | 19 | 12 | 16 | 15
  Leukocytes (/HPF): Many/TNTC: number analyzed (Participants) | 56 | 56 | 57 | 53
  Leukocytes (/HPF): Many/TNTC | 11 | 3 | 9 | 7
  Nitrite: Positive | 2 | 1 | 2 | 1
  Squamous Epithelial Cells (/HPF): Many/TNTC: number analyzed (Participants) | 54 | 54 | 54 | 49
  Squamous Epithelial Cells (/HPF): Many/TNTC | 6 | 0 | 6 | 8

9. Secondary Outcome: Number of Participants With Potentially Clinically Important Changes in Vital Signs and Body Weight
Description: Participant's vital signs and body weight were examined to determine the important changes. Vital signs included systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rate. mmHg= millimeters of mercury, DFB= Decrease from baseline and IFB= Increase from baseline.
Time Frame: From first dose of study drug administration (Day 1) up to 28 days after the last dose administration, 197 days
Population: The Safety analysis set included all participants who received at least 1 dose of the study drug post-randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PRV-015 100 mg | PRV-015 300 mg | PRV-015 600 mg
Number analyzed (Participants) | 57 | 56 | 57 | 54
Participants
  SBP: <=95 mmHg and DFB >=20 mmHg | 5 | 2 | 6 | 1
  SBP: >=160 mmHg and IFB >=20 mmHg | 2 | 1 | 0 | 1
  DBP: >=110 mmHg and IFB >=10 mmHg | 0 | 0 | 0 | 1
  Heart Rate: <=50 bpm and DFB >=20 bpm | 1 | 1 | 1 | 0
  Heart Rate: >=120 bpm and IFB >=20 bpm | 0 | 0 | 0 | 1
  Body weight: >=5% DFB | 8 | 11 | 9 | 7
  Body weight: >=5% IFB | 9 | 8 | 13 | 5

10. Secondary Outcome: Number of Participants With Anti-PRV-015 Antibodies
Description: Blood samples were collected to determine the presence of anti-drug antibodies by immunoassay.
Time Frame: Baseline (Day 1) and Weeks 2, 4, 12, 22, 24 and 28
Population: The Immunogenicity analysis set included participants who were randomized, dosed, and had at least 1 evaluable immunogenicity assessment. Only participants with data collected at specific time point are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | PRV-015 100 mg | PRV-015 300 mg | PRV-015 600 mg
Number analyzed (Participants) | 53 | 56 | 53
Participants
  Baseline: number analyzed (Participants) | 52 | 52 | 50
  Baseline | 3 | 8 | 7
  Week 2: number analyzed (Participants) | 53 | 56 | 51
  Week 2 | 8 | 9 | 9
  Week 4: number analyzed (Participants) | 52 | 51 | 48
  Week 4 | 5 | 6 | 5
  Week 12: number analyzed (Participants) | 51 | 51 | 53
  Week 12 | 4 | 5 | 4
  Week 22: number analyzed (Participants) | 49 | 49 | 48
  Week 22 | 4 | 4 | 2
  Week 24: number analyzed (Participants) | 49 | 51 | 49
  Week 24 | 4 | 3 | 2
  Week 28: number analyzed (Participants) | 50 | 52 | 48
  Week 28 | 4 | 3 | 2

11. Secondary Outcome: Minimum Serum Concentrations (Cmin) of PRV-015
Description: Blood samples were collected at specified timepoints to determine the Cmin.
Time Frame: Pre-dose on Day 1 and Weeks 2, 4, 8, 12, 16, 20, 22, 24 and 28
Population: The Pharmacokinetic (PK) analysis set included participants who were randomized, dosed, and had at least 1 post-dose evaluable PK assessment. Only participants with data collected at specific time point are reported. Participants were not analyzed at pre-dose on Day 1 as the study drug was not administered. Hence, no data collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | PRV-015 100 mg | PRV-015 300 mg | PRV-015 600 mg
Number analyzed (Participants) | 46 | 53 | 46
nanogram per milliliter
  Pre-dose on Day 1: number analyzed (Participants) | 0 | 0 | 0
  Week 2 | 8778 (74.1) | 27820 (39.8) | 66400 (46.1)
  Week 4: number analyzed (Participants) | 36 | 43 | 39
  Week 4 | 15140 (42.8) | 51190 (42.1) | 98420 (49.4)
  Week 8: number analyzed (Participants) | 31 | 40 | 33
  Week 8 | 21790 (46.4) | 61990 (66.5) | 142600 (43.7)
  Week 12: number analyzed (Participants) | 28 | 33 | 32
  Week 12 | 23630 (46.8) | 73150 (56.5) | 168300 (37.9)
  Week 16: number analyzed (Participants) | 25 | 27 | 26
  Week 16 | 22960 (46.7) | 75830 (65.1) | 166700 (44.9)
  Week 20: number analyzed (Participants) | 20 | 25 | 21
  Week 20 | 27000 (42.5) | 74110 (67.8) | 186400 (51.2)
  Week 22: number analyzed (Participants) | 20 | 22 | 21
  Week 22 | 25410 (36.2) | 73120 (64.2) | 181000 (55.6)
  Week 24: number analyzed (Participants) | 18 | 18 | 18
  Week 24 | 26680 (40.3) | 72400 (49.6) | 160500 (47.5)
  Week 28: number analyzed (Participants) | 26 | 25 | 27
  Week 28 | 10210 (58.0) | 32810 (80.0) | 69370 (78.3)

ADVERSE EVENTS:
Time Frame: Single-blind Period: From first dose of study drug administration (Day 1) up to 28 days. Double-blind Period: From first dose of study drug administration (Day 1) up to 28 days after the last dose administration, 197 days
Description: The Safety analysis set included all participants who received at least 1 dose of the study drug post-randomization.
Arm/Group | Single-blind: Placebo | Double-blind: Placebo | Double-blind: PRV-015 100 mg | Double-blind: PRV-015 300 mg | Double-blind: PRV-015 600 mg
All-Cause Mortality (participants affected / at risk) | 0/387 | 0/57 | 0/56 | 0/57 | 0/54
Serious Adverse Events (participants affected / at risk) | 2/387 | 1/57 | 0/56 | 0/57 | 1/54
Other Adverse Events (participants affected / at risk) | 0/387 | 22/57 | 18/56 | 22/57 | 19/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-blind: Placebo (N=387) | Double-blind: Placebo (N=57) | Double-blind: PRV-015 100 mg (N=56) | Double-blind: PRV-015 300 mg (N=57) | Double-blind: PRV-015 600 mg (N=54)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gluten Sensitivity (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single-blind: Placebo (N=387) | Double-blind: Placebo (N=57) | Double-blind: PRV-015 100 mg (N=56) | Double-blind: PRV-015 300 mg (N=57) | Double-blind: PRV-015 600 mg (N=54)
Covid-19 (Infections and infestations) | 0 (0) | 3 (3) | 5 (5) | 8 (8) | 5 (5)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 5 (6) | 3 (5) | 4 (4) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 4 (4) | 5 (5) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 6 (7) | 1 (1) | 4 (6) | 4 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 5 (5) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 3 (3) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 2 (2)
Injection Site Bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Injection Site Erythema (General disorders) | 0 (0) | 2 (2) | 3 (8) | 3 (6) | 2 (7)
Injection Site Reaction (General disorders) | 0 (0) | 1 (2) | 3 (4) | 3 (6) | 3 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/27/NCT04424927/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-17): https://cdn.clinicaltrials.gov/large-docs/27/NCT04424927/SAP_001.pdf